CLINICAL TRIAL: NCT04913402
Title: The Safety of Administration of Sufentanil by Paramedics to Treat Pain in Acute Trauma in The Prehospital Setting: Observational Study
Brief Title: Sufentanil Used by Paramedics to Treat Pain in Acute Trauma
Status: Completed | Type: Observational
Sponsor: Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O. (Other)
Collaborators: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Roman Sýkora, MD, Ph.D., Research coordinator, Zdravotnicka Zachranna Sluzba Karlovarskeho Kraje, P.O.
Other Study IDs: Sufentanil
Record Dates: First submitted 2021-05-17; First posted 2021-06-04 (Actual); Last update posted 2021-06-04 (Actual); Status verified 2021-05

CONDITIONS: Trauma Injury; Pain
Keywords: Sufentanil; Paramedic; Acute trauma injury; Prehospital emergency care
MeSH Terms: conditions — Accidental Injuries; Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Consultation: Patient who were administered sufentanil in acute trauma by paramedics after phone call consultation with medical doctor.
  Interventions: Other: Sufentanil administered by paramedics after the phone call consultation of medical doctor.
- Competency: Patient who were administered sufentanil in acute trauma by paramedics with competence to administer sufentanil without any consultation with medical doctor.
  Interventions: Other: Sufentanil administered by paramedics based on their competency, without consultation of medical doctor.

INTERVENTIONS:
Other: Sufentanil administered by paramedics after the phone call consultation of medical doctor. — Administration of sufentanil to patients with acute injury by paramedics only after phone-call consultation of medical doctor.
  Groups: Consultation
Other: Sufentanil administered by paramedics based on their competency, without consultation of medical doctor. — Administration of sufentanil to patients with acute injury by paramedics with competency to administer sufentanil without medical doctor consultation.
  Groups: Competency

SUMMARY:
The new competence of paramedics to administer opioid analgesics in acute trauma patients without presence or phone-call consult with an emergency medical doctor will be assessed in this study.

DETAILED DESCRIPTION:
The administration and indication of an opioid analgesics is carried by a medical doctor in most European emergency services. However, trips to majority of less serious traumas are realized by ambulances with paramedic crews without a medical doctor present on site. In this study will be assessed the new competence of paramedics to administer opioid analgesics without presence or phone-call consult with an emergency medical doctor.

This study will address the safety and efficacy of sufentanil administered by the paramedics in the field to patients with acute trauma without any consultation with medical doctors.

ELIGIBILITY:
Inclusion Criteria:

* acute trauma with severe pain (VAS/NRS > 4)
* age > 18 years
* conscious patient (GCS = 15; alert in AVPU)
* haemodynamically stable patient (> 100mmHg of systolic blood pressure, > 60/min of heart rate)

Exclusion Criteria:

* doctor on site
* paediatric patient
* predominantly chronic but not acute pain
* incomplete documentation
* other than traumatic reasons for opioid administration (eg. acute coronary syndrome)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults patient in prehospital emergency care, who suffered acute trauma with severe pain.
Sampling Method: Non-Probability Sample
Enrollment: 158 (Actual)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-03-23 (Actual); Study Completion 2021-05-15 (Actual)

PRIMARY OUTCOMES:
The safety of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - incidence of apnea | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - apnea - during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The safety of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - incidence of bradypnoea | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - bradypnoea - is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The safety of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - incidence of nausea. | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - nausea - is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The safety of pain treatment by the paramedics with competence to sufentanil administration in acute trauma - incidence of bradypnoea. | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of adverse effects of sufentanil administration in both study groups - vomiting - is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).
The efficacy of pain treatment by the paramedics with competence to sufentanil - administration in acute trauma - visual analogue scale. | Before sufentanil administration and at the handover of the patient to the hospital, up to 60 minutes.
  The ten point Visual analogue scale is used to measure the efficacy of pain treatment. The difference of VAS before administration of sufentanil and at the handover at the emergency department is calculated and compared in both groups (in points).
The efficacy of pain treatment by the paramedics with competence to sufentanil -administration in acute trauma - numeric rating scale. | Before sufentanil administration and at the handover of the patient to the hospital, up to 60 minutes.
  The ten point Numeric rating scale (NRS) is used to measure the efficacy of pain treatment. The difference of NRS before administration of sufentanil and at the handover at the emergency department is calculated and compared in both groups (in points).

SECONDARY OUTCOMES:
Dose of administered sufentanil | After sufentanil administration, up to 60 minutes.
  The average dose of administered sufentanil per each case (in micrograms) is reported in both groups.
Incidence of potentiation of analgesia by other analgesics | After sufentanil administration, up to 60 minutes.
  Number of cases of potentiation of analgesia by use of additional analgesics and is reported and compared in both groups (pertcentage).
Types of drugs used for potentiation of analgesia by sufentanil | After sufentanil administration, up to 60 minutes.
  The type and generic name of additional analgesics and is reported and compared in both groups (pertcentage).
The influence on haemodynamic parameters - non invasive blood pressure (BP) -systolic blood pressure | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of systolic blood pressure before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. Systolic blood pressure is measured in milimeters of hydrargyrum (mmHg).
The influence on haemodynamic parameters - non invasive blood pressure (BP) - diastolic blood pressure | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of diastolic blood pressure before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. Diastolic blood pressure is measured in milimeters of hydrargyrum (mmHg).
The influence on haemodynamic parameters - heart rate (HR) | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of heart rate before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. Heart rate is measured as monitored or palpated beats per minute (bpm).
The influence on peripheral oxygen saturation (SpO2) | Before sufentanil administration and at the time of the handover in hospital, up to 60 minutes.
  The difference of SpO2 before the administration of sufentanil and at the handover at the emergency department is measured, calculated and compared in both groups. SpO2 is measured as percentage.
Need for oxygenotherapy | After sufentanil administration up to the handover of the patient to the hospital, up to 60 minutes.
  Measurement of incidence of need for oxygenotherapy is measured during the period from sufentanil administration (baseline) up to handover of the patient to the hospital (percentage).

CONTACTS AND LOCATIONS:
Overall Officials: Roman SYKORA, PhD, Principal Investigator — Emergency Medical Service of Karlovy Vary Region, Czech Republic
Locations (1):
- Zdravotnická záchranná služba Karlovarského kraje, p.o., Karlovy Vary, Karlovarský kraj, Czechia

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request disposable by researchers.

REFERENCES:
- [Background] Gnirke A, Beckers SK, Gort S, Sommer A, Schroder H, Rossaint R, Felzen M. [Analgesia in the emergency medical service: comparison between tele-emergency physician and call back procedure with respect to application safety, effectiveness and tolerance]. Anaesthesist. 2019 Oct;68(10):665-675. doi: 10.1007/s00101-019-00661-0. Epub 2019 Sep 5. German. PMID 31489458
- [Result] Scharonow M, Alberding T, Oltmanns W, Weilbach C. Project for the introduction of prehospital analgesia with fentanyl and morphine administered by specially trained paramedics in a rural service area in Germany. J Pain Res. 2017 Nov 6;10:2595-2599. doi: 10.2147/JPR.S151077. eCollection 2017. PMID 29158691
- See also: website of Emergency Medical Service of Karlovy Vary Region — http://www.zzskvk.cz